NCT03923530

IRB 201901097

Pressure Assessment to Improve Outcomes after TAVR: a registry

## IRB 201901097 Pressure Assessment to Improve Outcomes after TAVR: a registry 5/14/2020

## NCT03923530

- 1.
- 2. We used Kolmogorov-Smirnov and Shapiro-wilk tests to examine distribution of our data. Despite small sample size, we had normal distribution. Therefore, we used parametrical approaches to compare means before and after the TAVR.
- 3. We used descriptive analysis to calculate Mean and standard deviation for age of the patients.
- 4. We used paired t-test to compare mean Kansas City Cardiomyopathy Questionnaire parameters, including physical limitation, symptom frequency, quality of life, social limitation, and overall summary before and after TAVR. We employed the paired t-test to compare mean of left ventricular end diastolic pressure, systolic and diastolic blood pressures before and after TAVR as well.
- 5. P value less than 0.05 was considered as statistically significant.
- 6. All statistics were done by SPSS software, version 24 (IBM Corp., Armonk, NY, USA).